CLINICAL TRIAL: NCT06526806
Title: The Effect of Use of Kahoot in Pediatric Emergency Nursing Course on Students' Course Success and Motivation Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Aslı Akdeniz Kudubeş, ASSOCIATE PROFESSOR, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AsliAkdenizKudubes
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Child, Only; Nurse's Role
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Students in the experimental group will be informed about the Kahoot game strategy. 1-7 and 9-15. After the end of each lesson in the following weeks (except the midterm exam week in the eighth week), students will play the "Kahoot" game consisting of a total of five questions for approximately 10 minutes in the classroom. The first five minutes will be planned as answering the questions, and the other five minutes will be planned as evaluating the results. Students' answers and score calculations will be automatically recorded in the system, allowing them to see correct and incorrect answers, and learning deficiencies will be identified.
  Interventions: Other: Kahoot game strategy
- Control group (No Intervention): The learning topics of the pediatric emergency nursing course will be conveyed to students through face-to-face education supported by PowerPoint presentations and learning methods such as video, question-answer-discussion. Kahoot game strategy will not be applied to students in the control group.

INTERVENTIONS:
Other: Kahoot game strategy — Students in the experimental group will be informed about the Kahoot game strategy. 1-7 and 9-15. After the end of each lesson in the following weeks (except the midterm exam week in the eighth week), students will play the "Kahoot" game consisting of a total of five questions for approximately 10 minutes in the classroom. The first five minutes will be planned as answering the questions, and the other five minutes will be planned as evaluating the results. Students' answers and score calculations will be automatically recorded in the system, allowing them to see correct and incorrect answers, and learning deficiencies will be identified. Measurements will be made with data collection tools in the first week, ninth (after the midterm exam) and eighteenth weeks (after the final exam) of the course.
  Other Names: education
  Arms: Experimental group

SUMMARY:
With the characteristics of the new generation and the innovations brought by the age, it has become inevitable to use new educational, instructive and entertaining methods in nursing education. Considering the problems experienced by nursing students with traditional education, the use of Kahoot will be a remarkable result in the literature. The gamification process with Kahoot encourages thinking skills in situations where the subject is sensitive and challenging, ensuring better retention of information and improving internal motivation. Therefore, in order to make learning efficient and to ensure the active participation of students, it should be processed using different interactive methods in nursing education. Pediatric emergency nursing course is a content-intensive and rich course that blends emergency and pediatric nursing, containing information on child health and development in addition to the learning outcomes of the emergency nursing course. This study was carried out within the scope of the pediatric emergency nursing course; It is thought that it will enable students to repeat the basic concepts of the course, master the terminology, and provide a supportive learning environment for pediatric emergency nursing, which is a difficult field for students, and will contribute to nursing education and nursing literature.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled study to determine the effect of using Kahoot in the pediatric emergency nursing course on students' course success and motivation levels.

ELIGIBILITY:
Inclusion Criteria:

* Those over 18 years of age,
* Third year nursing students,
* Taking the pediatric emergency nursing course for the first time,
* Those who have not experienced Kahoot before,
* Nursing students who volunteer to participate in the research will be included in the research.

Exclusion Criteria:

* Those who do not volunteer to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Exam score | Five months
  An increase in the exam score indicates an increase in the level of success.
Motivation Scale for Instructional Material mean scores | Five months
  An increase in the scale score indicates an increase in the motivation level.

CONTACTS AND LOCATIONS:
Overall Officials: ASLI KUDUBEŞ, Principal Investigator — BİLECİK ŞEYH EDEBALİ UNIVERSITY
Locations (1):
- Asli Kudubeş, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No